CLINICAL TRIAL: NCT05560984
Title: Cervical Internal os Plasty in Management of Placenta Previa and Focal Accreta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Al Shymaa Mohamed Abd El Hadi, Assistant lecturer,obstetrics and gynecology department, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cervix IO in placenta previa
Record Dates: First submitted 2022-09-24; First posted 2022-09-30 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Cervical IO Plasty in Management of Placenta Previa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study population (Experimental): Women with previous one or more cesarean sections with placenta previa and focal accrete
  Interventions: Combination Product: cervical internal os plasty

INTERVENTIONS:
Combination Product: cervical internal os plasty — A long Allis forceps will be passed through the uterine incision and used to grasp the anterior lip of the cervix, pulling the cervix upwards into the uterine cavity. An assistant sometimes needs to elevate the cervix upwards from the vaginal aspect. The anterior lip of the cervix will be sutured to the anterior wall of the lower uterine segment using two or three simple interrupted absorbable stitches (Vicryl or Vicryl rapid no. 0). This aids to compress the bleeding sites of the placental bed and support the very thin lower uterine segment. If the placenta was implanted posteriorly and the bleeding areas will be mainly from the posterior wall of the uterus, the same procedure could be repeated using the posterior lip of the cervix. A Hegar dilator (size 12) will be inserted in a retrograde manner from the abdominal aspect toensure patency of the cervical canal .

SUMMARY:
Aim of the work:

Better management & reducing hemorrhage and complication in patients placenta previa and focal accreta .

DETAILED DESCRIPTION:
Placenta accrete spectrum (PAS) is one of the major causes of massive obstetric hemorrhage and life-threatening complication of pregnancy. Patients with placenta previa may develop severe postpartum hemorrhage especially when coinciding with placenta accreta, it may be associated with potentially life-threatening maternal hemorrhage after removal of the placenta due to its incomplete separation and massive bleeding from the placental attachment site. Normally, the placenta adheres only to the decidua basalis, thus it separates smoothly from the wall of the uterus after delivery. Placenta accreta (PA) exists when the chorionic villi penetrate through the decidua basalis into the myometrium . The steady rise of cesarean section (CS) delivery rates in recent years combined with increasing maternal age, multiparity, placenta previa, prior uterine surgeries or curettage, and Asherman syndrome is associated with increasing incidence of PAS. In a systematic review, the rate of placenta accreta spectrum (PAS) increase from 0.3% in women with one previous cesarean delivery to 6.74% for women with five or more cesarean deliveries . In the setting of a placenta previa and one or more previous cesarean deliveries, the risk of PAS dramatically increases. For women with placenta previa, the risk of placenta accrete is 3%, 11%, 40%, 61%, 67%, for the first, second, third, fourth, and fifth or more cesareans, respectively. Placenta previa and placenta accrete carry significant maternal and fetal morbidity and mortality. The maternal mortality in women with PA may reach as high as 7-10 % . Acute torrential bleeding, massive blood transfusion, hysterectomy, and even the death of the woman can occur during cesarean delivery because of placenta previa increta. As intraoperative bleeding from PASin the lower uterine segment is often vast, massive, dramatically quick and difficult to stop after removal of the placenta resulting in severe maternal morbidity and mortality it is of outmost importance to have a pre-planned approach to this surgical challenge that is effective and swift. The differences between the lower and upper segments of the uterus are the main cause for postpartum hemorrhage associated with placenta accreta spectrum. The lower uterine segment is highly vascular and slower to retract than upper segment. Surgical intervention is indicated when uterotonic medications fail to control blood loss . The optimal management of PAS remains controversial. However, in practice, the conservative methods sometimes are incapable of stopping the bleeding from the placental attachment site. Moreover, the success of some surgical techniques, such as blood vessel ligation, has been associated with the experience and proficiency of the obstetricians, and in many hospitals, the conditions do not exist for performing perioperative temporary balloon occlusion of the internal iliac arteries and uterine arterial embolization. If these procedures prove invalid, hysterectomy is performed to ensure maternal survival. Currentseveral clinical hemostatic techniques have been described in the literature for controlling massive bleeding associated with placenta previa cesarean sections, including uterine packing with gauze , balloon tamponades,superposition sutures,hemostatic multiple square suturing, insertion of parallel vertical compression sutures , and so on when the bleeding is not so severe. If necessary, obstetricians often attempt to employ B-Lynch sutures, and embolization or ligation of the uterine and internal iliac arteries ,but there is a wide variation in the success rate of these maneuvers . There is lack of consensus on the optimal uterine sparing surgical approach to reduce intraoperative bleeding if the placenta is partially separated. Whilst electing for timely hysterectomy may be recommended and lifesaving, this may not be ideal for women wishing to preserve their fertility and uterine sparing alternative interventions are highly needed.

ELIGIBILITY:
Inclusion Criteria:

* All the participants with placent aprevia and focal accreta will be diagnosed by ultrasound and color Doppler.
* One or more previous cesarean section.
* Gestational age of 32 - 38 weeks.
* Desire to preserve the uterus

Exclusion Criteria:

* Diffuse placenta accreta.
* Placenta percreta.
* Presence of uncontrollable hemorrhage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
amount of intra-operative blood loss (mL) | 5 months

SECONDARY OUTCOMES:
Number of patients develop postpartum hemorrhage (500 mL or greater). | 5 months
Number of patients need blood transfusion | 5 months
Number of patients need hysterectomy | 5 months
Mean duration of postoperative hospital stay (days). | 5 months
Time needed to perform the technique (minutes). | 5 months
Number ot participants develop complications: •Urinary bladder injury •Wound infection •Postoperative fever. | 5 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauniaux E, Chantraine F, Silver RM, Langhoff-Roos J; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Epidemiology. Int J Gynaecol Obstet. 2018 Mar;140(3):265-273. doi: 10.1002/ijgo.12407. No abstract available. PMID 29405321
- [Background] Kondoh E. Expectant Management of Placenta Accreta Spectrum Disorders. Surg J (N Y). 2021 Jun 3;7(Suppl 1):S2-S6. doi: 10.1055/s-0040-1722240. eCollection 2021 Dec. PMID 35036541